CLINICAL TRIAL: NCT04616144
Title: Fresh Corneal Lenticule Implantation in Hyperopic Patients With High Astigmatism
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EHospitalP
Record Dates: First submitted 2020-10-26; First posted 2020-11-04 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Hyperopia; High Astigmatism
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Intervention Model Description: Miopic Group Hyperopic Group
Masking Description: Miopic Group Hyperopic Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FRESH CORNEAL LENTICULE IMPLANTATION (Other): The aim of this study is to investigate the effect of fresh corneal lenticule implantation as allogenic implant that will be taken from myopic patients to implant in hyperopic patients with high astigmatism using VisuMax Femtosecond Laser-Smile module surgery with primary objective to assess(increase) visual acuity (far, intermediate, near vision) and secondary objective to stabilize(decrease) high astigmatism by reducing K values. Fresh corneal lenticule implantation as allogenic implant that we took from myopic patients (-5.0D) to implant in hyperopic patients (+4.0 D +3.0cyl) according to high K2 values. The stromal pocket diameter was 8 mm, 4mm super incision and 130-µm cap thickness.
  Interventions: Device: Fresh Corneal Lenticule Implantation using Relex-Smile VisuMax Femtosecond Laser

INTERVENTIONS:
Device: Fresh Corneal Lenticule Implantation using Relex-Smile VisuMax Femtosecond Laser — Fresh Corneal Lenticule Implantation using ReLex-Smile

SUMMARY:
The refractive combination of high hyperopia with high astigmatism is difficult to treat surgically. In addition, there are not many suitable options to offer such patients presenting with this condition. The method used at the EYE Hospital Pristina using fresh lenticule implantation by ReLex-SMILE is safe and effective method. Fresh Corneal Implantation is a safe treatment for hyperopia with high astigmatism comparing with refractive IOL implantation (loss of accommodation, endophthalmitis). Its primary objective is to increase visual acuity, accommodation process, patient satisfaction which makes patient to enjoy a happier life. We believe this study will be the future of refractive surgery for treating high hyperopia.

DETAILED DESCRIPTION:
This study is to investigate the effect of fresh corneal lenticule implantation as allogenic implant that will be taken from myopic patients to implant in hyperopic patients with high astigmatism using VisuMax Femtosecond laser - Smile module surgery with primary objective to assess (increase) visual acuity (far, intermediate, near vision) and secondary objective to stabilize (decrease) high astigmatism by reducing K-values.

ELIGIBILITY:
Inclusion Criteria:

* patients with high spherical hyperopia over + 4.5 D
* astigmatism over + 3 cyl.
* corneal thickness minimum 450 µm and maximum 550 µm.

Exclusion Criteria:

* corneal thickness over 550 µm
* history of glaucoma
* retinal detachment
* cataract
* history of ocular inflammation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Increase of visual acuity, accommodation process | 12 months
  Using fresh myopic corneal lenticule resulted in the increase of the visual acuity (far, intermediate and near vision)

SECONDARY OUTCOMES:
Decrease of high hyperopic astigmatism | 12 months
  In order to stabilize high hyperopic astigmatism and reduce K-values, the myopic fresh corneal lenticule was implanted.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided